CLINICAL TRIAL: NCT02263053
Title: Immediate Effects of Posterior Mobilization Versus Caudal Mobilization in Patients With Temporomandibular Disorders: A Randomized Clinical Trial
Brief Title: Immediate Effects of Posterior Mobilization Versus Caudal Mobilization in Patients With Temporomandibular Disorders
Acronym: TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, Gabriel Peixoto Leão Almeida, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFCeara
Record Dates: First submitted 2014-09-26; First posted 2014-10-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posterior Mobilization (Active Comparator): Patient supine on the gurney, previously trained physiotherapist with disposable gloves, one hand place your thumb on the lower lateral incisors and canines. Applies a force previous distraction grade III and performs oscillating for 1 minute.
  Interventions: Procedure: CAUDAL MOBILIZATION
- Caudal Mobilization (Active Comparator): Patient supine on the gurney, previously trained physiotherapist with disposable gloves, one hand place your thumb on the lower molars of patients. Apply simultaneous flow and force the previous direction, and performs the degree of oscillation III for 1 minute.
  Interventions: Procedure: POSTERIOR MOBILIZATION

INTERVENTIONS:
Procedure: POSTERIOR MOBILIZATION — Patient supine on the gurney, previously trained physiotherapist with disposable gloves, one hand place your thumb on the lower lateral incisors and canines. Applies a force previous distraction grade III and performs oscillating for 1 minute.
  Arms: Caudal Mobilization
Procedure: CAUDAL MOBILIZATION — Patient supine on the gurney, previously trained physiotherapist with disposable gloves, one hand place your thumb on the lower molars of patients. Apply simultaneous flow and force the previous direction, and performs the degree of oscillation III for 1 minute.
  Arms: Posterior Mobilization

SUMMARY:
The Temporomandibular Joint (TMJ) is one of the most complex joints in the individual. It is composed of the mandibular condyle is positioned within the glenoid fossa of the temporal bone, and the articular disk that separates these two bones. The normal biomechanics of the TMJ is the concave / convex relationship between the condyles and the articular disc. The movements of the TMJ joint are: mandibular depression and elevation (opening and closing of the mouth), mandibular protrusion and retraction, and lateral deviations. The DTM is a musculoskeletal disorder of the masticatory system that affects over 25% of the population. Physical therapy can be adopted this treatment in order to relieve musculoskeletal pain, reduce inflammation and restore normal motor functions. The physical therapy interventions taken include electrotherapy, exercise therapy, acupuncture and manual therapy. Overall objective is to assess the immediate effects of previous mobilization versus flow amplitude of mandibular depression in patients with temporomandibular dysfunction. The type of study will be a randomized study of two parallel groups balanced distribution (1: 1) and double-blind. The research will be conducted in the Laboratory of Human Movement Analysis of Physiotherapy, Faculty of Medicine, Federal University of Ceará. The study population will consist of residents in the city of Fortaleza-CE individuals who voluntarily seek to participate in the study due to symptoms of TMD. Data, anthropometry, application of Research Diagnostic Criteria for Temporomandibular Disorders will be collected. The physiotherapist responsible for the assessment before and after the interventions will be blind with respect to the distribution of the treatment groups. The patient will also be blind, because you will not know whether or caudal anterior mobilization was performed. Randomization codes are generated by computer using Random Allocation Software (version 1.0.0) at a ratio of 1: 1 by a researcher not involved in the data collection. These codes will be placed in sealed, opaque envelopes being numbered consecutively, which will ensure the covert allocation of study participants. Our data are considered confidential as joint property of the parties involved.

ELIGIBILITY:
Inclusion Criteria:

* Individuals have not received the last 3 months treatment for TMD, who are not taking anti-inflammatory and / or analgesic for at least two weeks, you are not in the period of postoperative head and / or neck and to accept the participation in the study and signed the Instrument of Consent

Exclusion Criteria:

* Subjects with no teeth, history of metabolic diseases (such as hyper / hypothyroidism), neurological disorders, history of cancer in the last five years, active inflammatory arthritis, fractures, dislocations of the jaw or neck.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mandibular range of motion | Five minutes after mobilization
  The caliper is a measuring instrument that inform the millimetric values of mandibular depression, as measured the distance between the edges of the incisors of the maxilla and mandible. Three measurements of the active mouth opening will be held, where the individual experiencing pain, the measurement will be the beginning of it, if he does not feel pain, be gauged from the maximum amplitude of movement. Soon after the arithmetic mean of the measurements will be made.

SECONDARY OUTCOMES:
Pain Intensity | Five minutes after mobilization
  Numeric Ratig Scale for Pain - 0 (no pain) and 10 (worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel PL Almeida, MSc, Principal Investigator — Universidade Federal do Ceara
Locations (1):
- Federal University of Ceara, Fortaleza, Ceará, Brazil